CLINICAL TRIAL: NCT01286441
Title: A Randomized, Double-blind, Multi-center, Placebo-controlled, Dose-ranging, Efficacy and Safety Trial of a New Botanical Drug Product Containing East Indian Sandalwood Oil (EISO) for Treatment of Common Warts (Verruca Vulgaris)
Brief Title: A Trial of a Botanical Drug Containing East Indian Sandalwood Oil (EISO) for Treatment of Common Warts
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ViroXis Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIR001-01
Record Dates: First submitted 2011-01-27; First posted 2011-01-31 (Estimated); Results first posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Common Warts
Keywords: Verruca vulgaris
MeSH Terms: conditions — Warts

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo for East Indian Sandalwood Oil ointment administered topically twice daily
  Interventions: Drug: Placebo
- 10% EISO (Active Comparator): East Indian Sandalwood Oil ointment, 10% (w/w), applied topically twice daily
  Interventions: Drug: 10% EISO
- 20% EISO (Active Comparator): East Indian Sandalwood Oil ointment, 20% (w/w), applied topically twice daily
  Interventions: Drug: 20% EISO
- 30% EISO (Active Comparator): East Indian Sandalwood Oil ointment, 30% (w/w), applied topically twice daily
  Interventions: Drug: 30% EISO

INTERVENTIONS:
Drug: 10% EISO — During the Treatment Period, subjects will apply study medication (10% EISO) to all warts in the treatment area for 12 weeks and will then be followed for an additional 12 weeks. Subjects achieving complete resolution will continue to apply the study medication for the entire 12-week treatment period. During the Follow-up Period, subjects will be followed by telephone every 4 weeks for 12 weeks.
  Other Names: 10% East Indian sandalwood oil ointment
  Arms: 10% EISO
Drug: Placebo — During the Treatment Period, subjects will apply placebo to all warts in the treatment area for 12 weeks and will then be followed for an additional 12 weeks. Subjects achieving complete resolution will continue to apply the study medication for the entire 12-week treatment period. During the Follow-up Period, subjects will be followed by telephone every 4 weeks for 12 weeks.
  Other Names: sandalwood scented placebo ointment
  Arms: Placebo
Drug: 20% EISO — During the Treatment Period, subjects will apply study medication (20% EISO) to all warts in the treatment area for 12 weeks and will then be followed for an additional 12 weeks. Subjects achieving complete resolution will continue to apply the study medication for the entire 12-week treatment period. During the Follow-up Period, subjects will be followed by telephone every 4 weeks for 12 weeks.
  Other Names: 20% East Indian sandalwood oil ointment
  Arms: 20% EISO
Drug: 30% EISO — During the Treatment Period, subjects will apply study medication (30% EISO) to all warts in the treatment area for 12 weeks and will then be followed for an additional 12 weeks. Subjects achieving complete resolution will continue to apply the study medication for the entire 12-week treatment period. During the Follow-up Period, subjects will be followed by telephone every 4 weeks for 12 weeks.
  Other Names: 30% East Indian sandalwood oil Ointment
  Arms: 30% EISO

SUMMARY:
Nonclinical studies have shown sandalwood oil to have anti-inflammatory, anti-fungal, antiviral, and anti-bacterial activities. Previous clinical studies have shown East Indian Sandalwood oil to be promising as a treatment for common warts in adults and children.

The primary objective of this study is to evaluate the efficacy and safety of 10%, 20%, and 30% East Indian Sandalwood Oil (EISO) ointment compared with the ointment placebo administered twice daily (bid) for 12 weeks for the treatment of common warts (Verruca vulgaris).

ELIGIBILITY:
Inclusion Criteria:

1. Are male or female, and 18 years of age or older at enrollment;
2. Have 2 to 10 common warts (Verruca vulgaris) to be treated within a single 5 cm-by-5 cm contiguous area (the treatment area);
3. The treatment area can be located anywhere on the body except for the following prohibited areas: the eye area (including eyelids), lips, mouth cavity, nasal cavity, inner ear, palms of the hands, soles of the feet, or the anogenital area;
4. The total surface area of the warts to be treated is ≤600 mm2;
5. If female of childbearing potential, have a negative urine pregnancy test at Screening and Randomization/Day 1, and are willing to use effective contraception during the study (ie, oral, implanted, or injectable contraceptives, intrauterine device (IUD), diaphragm, condom, tubal ligation, abstinence, or are in a monogamous relationship with a partner who has had a vasectomy);
6. Are judged to be in good health based upon the results of a physical examination, medical history, and safety laboratory tests;
7. Are willing and able to provide written informed consent;
8. Agree to use no wart-removing product (prescription or over-the-counter [OTC]) other than the study product during the course of the study;
9. Are willing and able to comply with the requirements of the study;
10. Are free of any systemic or dermatologic disorder, which, in the opinion of the investigator, will interfere with the study results or increase the risk of AEs.
11. Are willing to refrain from using cosmetics or other topical products in the treatment area for the duration of the study.

Exclusion Criteria:

1. Have less than 2 or more than 10 common warts within the designated treatment area;
2. Have warts outside of the treatment area that would interfere with study procedures or analyses;
3. Have participated in an investigational trial within 30 days prior to enrollment;
4. Have participated in a prior trial investigating EISO use for the treatment of common warts;
5. Have used salicylic acid or any over-the-counter wart-removing product in the treatment area within 30 days prior to enrollment;
6. Have used or will use oral zinc and/or cimetidine within 30 days prior to enrollment or during the course of the study;
7. Have received cryotherapy in the treatment area within 60 days prior to enrollment;
8. Have required or will require systemic intake of immunosuppressive or immunomodulatory medication (including oral or parenteral corticosteroids) within 30 days prior to enrollment or during the course of the study. Routine use of inhaled or intranasal corticosteroids during the study is allowed;
9. Have any current and/or recurrent pathologically relevant skin infections in the treatment area other than common warts (with the exception of Herpes simplex virus labialis);
10. Have any current uncontrolled infection;
11. Are pregnant, plan to become pregnant, or are breastfeeding;
12. Have a known sensitivity to any of the constituents of the investigational or control products including sandalwood oil, fragrances, or any members of the Compositae family of vascular plants (eg, sunflowers, daisies, dahlias, etc.);
13. Have any chronic or acute medical condition that, in the opinion of the investigator, may interfere with the study results or place the subject at undue risk (including human immunodeficiency virus, systemic lupus erythematosis, viral hepatitis, etc.);
14. Have any active malignancy or are undergoing treatment for any malignancy other than nonmelanoma skin cancer;
15. Have, in the opinion of the investigator, clinically significant clinical laboratory results at the time of screening that may interfere with the study results or place the subject at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2012-11; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Rogers, Arkansas
  - Fremont, California
  - Lomita, California
  - Miami, Florida
  - Arlington Heights, Illinois
  - Elwood, Indiana
  - Owensboro, Kentucky
  - Beverly, Massachusetts
  - Haverhill, Massachusetts
  - Fort Gratiot, Michigan
  - Newington, New Hampshire
  - Portsmouth, New Hampshire
  - Rochester, New York
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Columbus, Ohio
  - College Station, Texas
  - Dallas, Texas
  - San Antonio, Texas
  - Virginia Beach, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | 10% EISO | 20% EISO | 30% EISO
Started | 45 | 44 | 46 | 48
Completed | 38 | 37 | 39 | 37
Not Completed | 7 | 7 | 7 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 10% EISO | 20% EISO | 30% EISO | Total
Number analyzed (Participants) | 45 | 44 | 46 | 48 | 183
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (15.4) | 43.2 (17.5) | 44.3 (17.9) | 39.5 (15.2) | 43.3 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 24 | 27 | 28 | 105
  Male | 19 | 20 | 19 | 20 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 15 | 14 | 13 | 55
  Not Hispanic or Latino | 32 | 29 | 32 | 35 | 128
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 0 | 3 | 1 | 3 | 7
  White | 44 | 39 | 43 | 41 | 167
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 45 | 44 | 46 | 48 | 183
Height [Mean (Standard Deviation); unit: cm] | 165.2 (18.7) | 167.8 (9.9) | 167.5 (11.1) | 168.1 (10.5) | 167.2 (13.0)
Weight [Mean (Standard Deviation); unit: kg] | 81.8 (21.3) | 79.0 (18.1) | 75.9 (17.4) | 77.8 (20.5) | 78.6 (19.4)

OUTCOME MEASURES:

1. Primary Outcome: Complete Resolution of All Treated Warts by or at Week 12
Description: During the Treatment Period, subjects will apply study medication to all warts in the treatment area for 12 weeks and will then be followed for an additional 12 weeks. Subjects achieving complete resolution will continue to apply the study medication for the entire 12-week treatment period. During the Follow-up Period, subjects will be followed by telephone every 4 weeks for 12 weeks. Clinical evaluations, including wart counts, wart measurements and recording of adverse events and concomitant medications will be performed. Photographs of the treatment area will be taken at all study visits
Time Frame: 12 weeks
Population: FAS population was used for this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 10% EISO | 20% EISO | 30% EISO
Number analyzed (Participants) | 43 | 42 | 45 | 43
Participants | 2 | 5 | 2 | 3

2. Secondary Outcome: Number of Subjects Achieving Partial Resolution of Treated Warts
Description: Partial Resolution is defined as >/= 75% Reduction of treated wart
Time Frame: 12 weeks
Population: FAS population used for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 10% EISO | 20% EISO | 30% EISO
Number analyzed (Participants) | 43 | 42 | 45 | 43
Participants | 2 | 4 | 5 | 8

ADVERSE EVENTS:
Time Frame: Over the entire duration of the treatment and follow up periods (24 WEEKS)
Arm/Group | Placebo | 10% EISO | 20% EISO | 30% EISO
Serious Adverse Events (participants affected / at risk) | 0/45 | 1/44 | 0/46 | 0/48
Other Adverse Events (participants affected / at risk) | 3/45 | 0/44 | 0/46 | 3/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=45) | 10% EISO (N=44) | 20% EISO (N=46) | 30% EISO (N=48)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=45) | 10% EISO (N=44) | 20% EISO (N=46) | 30% EISO (N=48)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Application Site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less